CLINICAL TRIAL: NCT03010579
Title: Efficacy and Safety of Erythropoietin in the Treatment of Anemia in Patients With Lymphoma After Autologous Hematopoietic Stem Cell Transplantation
Brief Title: Erythropoietin in the Treatment of Anemia After Autologous Hematopoietic Stem Cell Transplantation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Jun Zhu, Chairman of Lymphoma Department, Peking University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKU-2016KT64
Record Dates: First submitted 2016-12-29; First posted 2017-01-05 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Anemia; Lymphoma; Hematopoietic Stem Cell Transplantation
Keywords: Anemia; Lymphoma; Hematopoietic stem cell transplantation; Erythropoietin
MeSH Terms: conditions — Anemia; Lymphoma | interventions — Erythropoietin; Hematinics; ferrous succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- erythropoietin group (Experimental): For those lymphoma patients with hemoglobin level less than 100 g/L on day +15 after autologous hematopoietic stem cell transplantation, erythropoietin will be administered. If necessary,oral ferrous succinate vitamins B12 and folic acid will be administered.
  Interventions: Drug: erythropoietin
- iron supplementation (Active Comparator): If necessary，oral ferrous succinate, vitamins B12 and folic acid will be administered.
  Interventions: Drug: iron supplementation

INTERVENTIONS:
Drug: erythropoietin — Erythropoietin will be administered subcutaneously (s.c.) at the dose of 10 000 IU, three times a week. If necessary,oral ferrous succinate vitamins B12 and folic acid will be administered.
  Other Names: Erythropoiesis-Stimulating Agent
  Arms: erythropoietin group
Drug: iron supplementation — If necessary, oral ferrous succinate, vitamins B12 and folic acid will be administered.
  Other Names: ferrous succinate
  Arms: iron supplementation

SUMMARY:
This is an randomized trial to evaluate the potential benefit of erythropoietin in the treatment of anemia in patients with lymphoma after autologous hematopoietic stem cell transplantation.

DETAILED DESCRIPTION:
Lymphoma patients with anemia on day +15 post-transplant will be randomized to erythropoietin group or control group. Potential benefit of erythropoietin will be evaluatedon day +60 post-transplant.

ELIGIBILITY:
Inclusion Criteria:

* confirmed lymphoma
* first autologous hematopoietic stem cell transplantation
* hemoglobin level less than 100 g/L on day +15 post-transplant
* written informed consent given by patient or his/her guardian if of minor age.

Exclusion Criteria:

* HIV positive
* Known allergy to recombinant human erythropoietin
* Uncontrolled infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
complete hemoglobin response rate | from day +15 to day +60 after autologous hematopoietic stem cell transplantation
  proportion of complete correctors (reaching hemoglobin 120 g/L in male patients, 110 g/L in female patients) before day +60 post-transplant

SECONDARY OUTCOMES:
proportion of participants with red blood cell transfusions | from day +15 to day +60 after autologous hematopoietic stem cell transplantation
  proportion of participants with red blood cell transfusions from day +15 to day +60 post-transplant
proportion of participants with deep vein thrombosis | from day +15 to day +60 after autologous hematopoietic stem cell transplantation
  proportion of participants with deep vein thrombosis from day +15 to day +60 post-transplant

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital & Institute, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No